CLINICAL TRIAL: NCT05292755
Title: Effects of Carboxymethylcellulose Artificial Tears on the Eye Microbiome: a Randomized, Controlled, Double-Blind Study
Brief Title: Effects of Carboxymethylcellulose Artificial Tears on the Eye Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202200427 -A
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium; MCC protocol; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Carboxymethylcellulose (CMC) Artificial Tears (Experimental): Refresh brand artificial tears containing 0.5% carboxymethylcellulose will be self-administered three times a day in each eye by the participants for 1 week in the experimental arm.
  Interventions: Drug: Carboxymethylcellulose (CMC) Artificial Tears
- Preservative-free, CMC-free Artificial Tears (Placebo Comparator): Systane brand artificial tears containing 0.4% polyethylene glycol 400 and 0.3% propylene glycol will be self-administered three times a day in each eye by the participants for 1 week in the control arm.
  Interventions: Drug: Preservative-free, CMC-free Artificial Tears (control)

INTERVENTIONS:
Drug: Carboxymethylcellulose (CMC) Artificial Tears — A pack of 21 vials of artificial tears containing carboxymethylcellulose 0.5% will be given to subjects in the treatment group.
  Other Names: Refresh Plus
  Arms: Carboxymethylcellulose (CMC) Artificial Tears
Drug: Preservative-free, CMC-free Artificial Tears (control) — A pack of 21 vials of artificial tears containing 0.4% polyethylene glycol 400 and 0.3% propylene glycol will be given to subjects in the control group.
  Other Names: Systane Ultra PF
  Arms: Preservative-free, CMC-free Artificial Tears

SUMMARY:
Carboxymethylcellulose (CMC), a common component in artificial tears, has been shown to modify the gut microbiome. The study is examining its effects on the eye microbiome, which may have implications on ocular disease and artificial tear choice. The study will administer artificial tears containing CMC to the treatment group and artificial tears without CMC to the control group. Surveys and conjunctival swabs will be collected before and after treatment for bacterial genome sequencing and analyzed by R statistical packages.

ELIGIBILITY:
Inclusion Criteria:

* Adults above age 18 of either sex who can self-administer artificial tears and return for follow-up at the UF Oaks Eye Clinic.

Exclusion Criteria:

* Individuals with active eye infections or have prosthetic eyes.
* Are immunocompromised, or are diagnosed with autoimmune diseases or malignant neoplasms about the eye.
* Individuals who take immunomodulatory therapy, steroids, antibiotics, medicated eyedrops, or are already using CMC eyedrops within 1 week of the study will also be excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yujia Zhou, Principal Investigator — University of Florida
Locations (1):
- University of Florida Oaks Eye Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou Y, Sidhu GS, Whitlock JA, Abdelmalik B, Mayer Z, Li Y, Wang GP, Steigleman WA. Effects of Carboxymethylcellulose Artificial Tears on Ocular Surface Microbiome Diversity and Composition, A Randomized Controlled Trial. Transl Vis Sci Technol. 2023 Aug 1;12(8):5. doi: 10.1167/tvst.12.8.5. PMID 37555738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Started | 40 | 40
Completed | 35 | 31
Not Completed | 5 | 9
Not completed — Lost to Follow-up | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (17.4) | 40.2 (13.8) | 40.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 13 | 12 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80
Contact lens use [Count of Participants; unit: Participants] | 9 | 10 | 19
Ocular surgery history [Count of Participants; unit: Participants] | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Species Richness
Description: Sampled 16S rRNA sequences were organized into 'operational taxonomic units' (OTUs) at a 97% sequence similarity threshold, and a phylogenetic tree was constructed from sampled OTUs using the QIIME2 bioinformatics platform. Faith's phylogenetic diversity was used as a measure of species richness, calculated as the sum of all phylogenetic tree branch lengths using the QIIME2 faith_pd plugin. The units for this measure are the number of nucleotide substitutions (phylogenetic distance, i.e. length) per branch, which is a scale measure from zero to infinity. Zero indicates a completely homogenous sample, and higher scores indicate greater species richness.
Time Frame: Assessed at day 1 and day 7, day 7 reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
units on a scale | 11.0 (2.1) | 11.1 (3.3)
Statistical Analysis 1: Comparison: Carboxymethylcellulose (CMC) Artificial Tears vs Preservative-free, CMC-free Artificial Tears; Test type: Other — One-way ANOVA was used to compare mean Faith's phylogenetic diversity before and after treatment for each intervention group at a two-tailed 95% confidence interval; p = 0.232, ANOVA

2. Primary Outcome: Species Diversity
Description: Sampled 16S rRNA sequences were organized into 'operational taxonomic units' (OTUs) at a 97% sequence similarity threshold. Shannon's diversity index was used as a measure of species diversity, calculated as the sum of -p/ln(p), where p is the proportion of the sample made up of each OTU using the QIIME2 shannon_pd plugin. This measure is a unitless scale proportion ranging from zero to infinity. Zero indicates a completely homogenous sample, and higher scores indicate greater species diversity.
Time Frame: Assessed at day 1 and day 7, day 7 reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
score on a scale | 3.9 (1.1) | 4.1 (1.1)
Statistical Analysis 1: Comparison: Carboxymethylcellulose (CMC) Artificial Tears vs Preservative-free, CMC-free Artificial Tears; ANOVA was used to compare mean Shannon's diversity indices before and after treatment for each intervention group at a two-tailed 95% confidence interval; Test type: Other; p = 0.224, ANOVA

3. Primary Outcome: Beta Diversity (Unweighted UniFrac)
Description: Sampled 16S rRNA sequences were organized into 'operational taxonomic units' (OTUs) at a 97% sequence similarity threshold, and a phylogenetic tree was constructed from sampled OTUs using the QIIME2 bioinformatics platform. Unweighted UniFrac distances were calculated as the number of shared nucleotide substitutions between two samples divided by the number of shared nucleotide substitutions among all samples using the QIIME2 unifrac plugin. The unweighted UniFrac is a unitless scale proportion ranging from zero to one. Greater UniFrac distances indicate greater beta diversity.
Time Frame: Assessed at day 1 and day 7, difference between day 1 and day 7 reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
score on a scale | 0.482 [0.388 to 0.574] | 0.529 [0.417 to 0.618]
Statistical Analysis 1: Comparison: Carboxymethylcellulose (CMC) Artificial Tears vs Preservative-free, CMC-free Artificial Tears; Repeated measures Mann-U-Whitney tests were used to compare changes in weighted and unweighted UniFrac distances between intervention groups before and after intervention at a two-tailed 95% confidence interval; Test type: Other; p = 0.227, Repeated measures Mann-U-Whitney

4. Primary Outcome: Beta Diversity (Weighted UniFrac)
Description: Sampled 16S rRNA sequences were organized into 'operational taxonomic units' (OTUs) at a 97% sequence similarity threshold, and a phylogenetic tree was constructed from sampled OTUs using the QIIME2 bioinformatics platform. Weighted UniFrac distances were calculated as the number of shared nucleotide substitutions between two samples divided by the number of shared nucleotide substitutions among all samples using the QIIME2 unifrac plugin, with samples weighted by abundance of species. The weighted UniFrac (weighted by number of duplicate OTUs) is a unitless scale proportion ranging from zero to infinity. Greater UniFrac distances indicate greater beta diversity.
Time Frame: Assessed at day 1 and day 7, difference between day 1 and day 7 reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
score on a scale | 0.584 [0.416 to 0.839] | 0.593 [0.468 to 0.797]

5. Secondary Outcome: Ocular Surface Disease Index Score
Description: The Ocular Surface Disease Index (OSDI) is a 12-item scale for the assessment of symptoms related to dry eye disease and their effect on vision. Participants conducted a survey before and after intervention, and the difference will be used as the outcome measure. The OSDI ranges from 0 to 48, and a higher score indicates greater ocular surface dryness. If reporting the difference, a more negative change in OSDI indicates greater improvement in dry eye symptoms. Pairwise Wilcoxon signed rank tests were used to compare changes in OSDI between intervention groups at a two-tailed 95% confidence interval.
Time Frame: Assessed at day 1 and day 7, difference between day 1 and day 7 reported.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
score on a scale | -1 [-5.5 to 0] | -2 [-4 to 0]

6. Secondary Outcome: Artificial Tear Use
Description: Patients will be asked 1 week after intervention how many times they administered eye drops each day. This measures compliance with intervention, ranging from zero drops per day to infinite drops per day. If a patient is perfectly compliant, the number of drops should be 3. Mann-U-Whitney tests were used to compare compliance between intervention groups at a two-tailed 95% confidence interval.
Time Frame: Assessed at day 7
Measure: Mean (Standard Deviation); unit: eyedrops per day
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
Number analyzed (Participants) | 35 | 31
eyedrops per day | 2.86 (0.81) | 2.16 (0.82)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for a duration of 7 days, from start of intervention to end of intervention 7 days after start of intervention.
Arm/Group | Carboxymethylcellulose (CMC) Artificial Tears | Preservative-free, CMC-free Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT05292755/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT05292755/ICF_001.pdf